CLINICAL TRIAL: NCT00428103
Title: Destiny Trial: Effects of Mitral Valve Annuloplasty With the Geoform Ring on Left Ventricular Geometry and Function in Patients With Cardiomyopathy
Brief Title: Effects of Mitral Valve Repair With the Geoform Ring on Cardiomyopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Crestanello, MD (Other)
Collaborators: Edwards Lifesciences (Industry); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Juan Crestanello, MD, Associate Professor of Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006H0138; 0006378 (Other: OSU surgery dept)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Mitral Valve Regurgitation; Congestive Heart Failure; Cardiomyopathy
Keywords: Mitral valve regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: 3 dimensional echocardiography — Lab tests: BNP, 6 minute walk test Transthoracic 3D echocardiogram

SUMMARY:
The primary aim of this study is to assess the changes on the shape and function of the left ventricle in patients with severe mitral valve regurgitation due to congestive heart failure and cardiomyopathy who undergo mitral valve reconstruction with a Geoform ring. Three-dimensional echocardiogram will be used for precise evaluation of the shape and function of the ventricle.

DETAILED DESCRIPTION:
Congestive heart failure is a leading cause of hospitalization and mortality with an estimated 5 million people affected in the United States of America. Ischemic and idiopathic (dilated) cardiomyopathies are the two most common etiologies. As the left ventricle fails, changes in ventricular geometry and function occurs that leads to functional mitral regurgitation. Mitral regurgitation is a complication of end stage cardiomyopathy that adversely affects survival and patient's functional status. Mitral regurgitation in these patients is not an intrinsic disease of the mitral valve but rather results from mitral annular dilatation and ventricular dilatation.

Geoform mitral annuloplasty ring reduces the antero-posterior diameter of the mitral valve and elevates the posterior mitral annulus. Although it has been very effective on eliminating mitral regurgitation its effects on ventricular geometry have not been fully elucidated. Evaluation of ventricular and mitral valve geometry and function and their interactions has been difficult. The availability of three dimensional echocardiogram with sophisticated finite volume analysis allows us to evaluate the changes in ventricular geometry associated with the implantation of the Geoform ring. We have then designed this study with the purpose of evaluating the changes in left ventricular geometry and function resulting from mitral valve annuloplasty with the Geoform ring in patients with left ventricular dysfunction and congestive heart failure.

The two primary endpoints of this study will be:

1. To assess the changes on left ventricular geometry and function as assessed by 3D echocardiography in patients with cardiomyopathy and severe mitral regurgitation who undergo mitral valve annuloplasty with a Geoform ring. This assessment will be done preoperatively, at three months, at six months, at one year, and at two years after the procedure.
2. To evaluate the effects on mitral valve annuloplasty with a Geoform ring on functional status.

   Secondary endpoints will be:
3. To evaluate the effect of mitral valve annuloplasty with a Geoform ring on mortality.
4. To evaluate its effects on hospitalization for congestive heart failure.
5. To evaluate the effect on the need of further interventions for congestive heart failure (insertion of ventricular assist device, transplantation, cardiac resynchronization therapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients would be at least 18 years old.
* They will have history of congestive heart failure and be in New York Heart Association Class III or IV.
* Their left ventricular ejection fraction will be less or equal to 30%.
* They will have moderate or severe mitral regurgitation as determined by echocardiogram. Echocardiogram's criteria for severe mitral regurgitation will be:

  * regurgitant volume greater than 50 ml,
  * regurgitant fraction greater than 50% and
  * effective regurgitant orifice greater than 40 mm2.

If the quantitative criteria are not available, severity of the MR will be graded qualitative in grades I, II, III, and IV. Patients with mitral regurgitation in grade III and IV will be eligible to be included in the study.

Exclusion Criteria:

* Cancer - Metastatic or any cancer within five years except patients with non- melanoma skin cancer.
* Recent stroke (less than six months).
* Severe COPD (patients with an FEV1 less than .8 liters).
* Patients on inotropic infusion preoperatively.
* Patients in atrial fibrillation.
* Pregnant patients.
* Patients with any other valvular disease that required surgical intervention except tricuspid valve disease.
* Patients that will require surgical ventricular restoration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To assess changes on left ventricular geometry and function using 3D echocardiography in patients with cardiomyopathy and severe mitral regurgitation who undergo mitral valve annuloplasty with a Geoform ring. | Post operative Mitral Valve repair
To evaluate effects on mitral valve annuloplasty with a Geoform ring on functional status. | Postoperative Mitral Valve repair

SECONDARY OUTCOMES:
To evaluate effect of mitral valve annuloplasty with a Geoform ring on mortality. | Postoperative
To evaluate effects on hospitalization for congestive heart failure. | Hospital admissions that occur after intial postoperative discharge
To evaluate effect on the need of further interventions for congestive heart failure (insertion of ventricular assist device, transplantation, cardiac resynchronization therapy). | Postoperative Mitral Valve repair

CONTACTS AND LOCATIONS:
Overall Officials: Juan Crestanello, MD, Principal Investigator — Ohio State University; Nadia Nathan, MD, Principal Investigator — Ohio State University; Subha Raman, MD, Principal Investigator — Ohio State University; Steven Bolling, MD, Principal Investigator — University of Michigan; Min Pu, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Smolens IA, Bolling SF. Surgical approaches to dilated cardiomyopathy. Curr Cardiol Rep. 2000 Mar;2(2):99-105. doi: 10.1007/s11886-000-0005-6. PMID 10980879
- [Background] Romano MA, Bolling SF. Update on mitral repair in dilated cardiomyopathy. J Card Surg. 2004 Sep-Oct;19(5):396-400. doi: 10.1111/j.0886-0440.2004.04079.x. PMID 15383049
- [Background] Levi GS, Bolling SF, Bach DS. Eccentric mitral regurgitation jets among patients having sustained inferior wall myocardial infarction. Echocardiography. 2001 Feb;18(2):97-103. doi: 10.1046/j.1540-8175.2001.00097.x. PMID 11262532
- [Background] Romano MA, Bolling SF. Mitral valve repair as an alternative treatment for heart failure patients. Heart Fail Monit. 2003;4(1):7-12. PMID 12808479
- [Background] Badhwar V, Bolling SF. Mitral valve surgery in the patient with left ventricular dysfunction. Semin Thorac Cardiovasc Surg. 2002 Apr;14(2):133-6. doi: 10.1053/stcs.2002.32314. PMID 11988951
- [Background] Bolling SF. Mitral reconstruction in cardiomyopathy. J Heart Valve Dis. 2002 Jan;11 Suppl 1:S26-31. PMID 11843517
- [Background] Bolling SF, Smolens IA, Pagani FD. Surgical alternatives for heart failure. J Heart Lung Transplant. 2001 Jul;20(7):729-33. doi: 10.1016/s1053-2498(01)00239-x. PMID 11448798
- [Background] Smolens IA, Pagani FD, Bolling SF. Mitral valve repair in heart failure. Eur J Heart Fail. 2000 Dec;2(4):365-71. doi: 10.1016/s1388-9842(00)00125-2. PMID 11113712
- [Background] Bolling SF. Mitral valve reconstruction in the patient with heart failure. Heart Fail Rev. 2001 Sep;6(3):177-85. doi: 10.1023/a:1011421014480. PMID 11391035
- [Background] Otsuji Y, Handschumacher MD, Schwammenthal E, Jiang L, Song JK, Guerrero JL, Vlahakes GJ, Levine RA. Insights from three-dimensional echocardiography into the mechanism of functional mitral regurgitation: direct in vivo demonstration of altered leaflet tethering geometry. Circulation. 1997 Sep 16;96(6):1999-2008. doi: 10.1161/01.cir.96.6.1999. PMID 9323092
- [Background] Verhey JF, Nathan NS, Rienhoff O, Kikinis R, Rakebrandt F, D'Ambra MN. Finite-element-method (FEM) model generation of time-resolved 3D echocardiographic geometry data for mitral-valve volumetry. Biomed Eng Online. 2006 Mar 3;5:17. doi: 10.1186/1475-925X-5-17. PMID 16512925